CLINICAL TRIAL: NCT01013259
Title: Explorative Analysis of the Immunomodulatory Capacities of Apathogenic Escherichia Coli Nissle 1917 in Patients With Rhinoconjunctivitis Due to Grass Pollen Allergy
Brief Title: Immunomodulation of E.Coli Nissle 1917 in Patients With Grass Pollen Rhinoconjunctivitis
Acronym: Ecorhino
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Prof. Dr. med. Margitta Worm, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ecorhino
Record Dates: First submitted 2009-11-10; First posted 2009-11-13 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Rhinoconjunctivitis
Keywords: E.coli; Mutaflor; grass pollen; rhinoconjunctivitis; rhinoconjunctivitis caused by grass pollen
MeSH Terms: conditions — Escherichia coli Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Mutaflor (Experimental)
  Interventions: Drug: Mutaflor

INTERVENTIONS:
Drug: Mutaflor — 1 capsule contains 2.5 - 25 billion viable bacteria of the strain E. coli Nissle 1917, 1 capsule daily over the first 4 days, 2 capsules daily until the end of treatment
  Arms: Mutaflor
Drug: Placebo — 1 placebo capsule matching the experimental treatment, according to the experimental arm
  Arms: Placebo

SUMMARY:
Due to the worldwide increasing prevalence of the allergic rhinoconjunctivitis, new therapeutical strategies are needed. The symptomatic treatment with topical and systemic antihistamines and corticosteroids are often insufficient. E.coli Nissle 1917 has immunomodulatory capacities and reveals less side effects. E.coli Nissle 1917 has no sedative properties and exhibits no hepatotoxic qualities. Thus, E.coli Nissle 1917 represents a new relevant therapeutical agent.

ELIGIBILITY:
Inclusion Criteria:

* clinical relevant grass pollen allergy with required treatment since 2 years
* positive skin prick test to grass
* positive sIgE towards grass (CAP 2)
* written informed consent

Exclusion Criteria:

* perennial rhinoconjunctivitis
* sinusitis
* chronic diarrhoea and other existing severe gastrointestinal diseases
* current specific immunotherapy to grass pollen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-02; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
symptom-medication score | 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Margitta Worm, Prof. Dr. med., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany